CLINICAL TRIAL: NCT03402152
Title: Validation of the Glx Biomarker for Treatment of Moderate Bipolar Depression With NRX-101
Brief Title: NRX101 Glx Biomarker Validation Study
Acronym: NRX-GLX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NeuroRx, Inc. (Industry)
Collaborators: Target Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRX101_004; NCT03401164 (obsolete NCT alias)
Record Dates: First submitted 2018-01-04; First posted 2018-01-18 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Bipolar Depression; Suicidal Ideation
Keywords: Biomarker
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and Care Providers will be masked with regard to medication administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRX-101 vs. Placebo (Experimental): Following study enrollment and randomization, subjects will undergo two treatment sessions, 3 days apart. Each treatment session will be conducted while the subject is undergoing Magnetic Resonance Spectroscopy to measure Glx in the ACC. In one treatment session the subject will receive oral placebo and in the other treatment session the subject will receive oral NRX-101. Following the second treatment session, the subject will participate in a four week open study of NRX-101, at the end of which a third session of Magnetic Resonance Spectroscopy will be conducted.
  Interventions: Drug: NRX-101; Drug: Placebo
- NRX-101 vs. lurasidone HCl (Experimental): Following study enrollment and randomization, subjects will undergo two treatment sessions, 3 days apart. Each treatment session will be conducted while the subject is undergoing Magnetic Resonance Spectroscopy to measure Glx in the ACC. In one treatment session the subject will receive oral lurasidone and in the other treatment session the subject will receive oral NRX-101. Following the second treatment session, the subject will participate in a four week open study of NRX-101, at the end of which a third session of Magnetic Resonance Spectroscopy will be conducted.
  Interventions: Drug: NRX-101; Drug: Lurasidone HCl

INTERVENTIONS:
Drug: NRX-101 — NRX-101, a fixed dose combination of D-cycloserine+lurasidone will be given twice a day by mouth
Drug: Lurasidone HCl — Lurasidone HCl will be given twice a day by mouth
  Arms: NRX-101 vs. lurasidone HCl
Drug: Placebo — Placebo oral capsule
  Arms: NRX-101 vs. Placebo

SUMMARY:
Subnormal level of Glutamate+Glutamine (Glx) in the Anterior Cingulate Cortex (ACC) of the brain has been associated with depression and PTSD. Similarly, interventions that increase the level of Glx in the brain, specifically electroconvulsive therapy (ECT) and intravenous ketamine infusion have been associated with a rapid decrease in depression and suicidal ideation. This effect has been demonstrated in a dose-dependent manner in randomized clinical assessments. D-cycloserine, a glycine site modulator of NMDA receptor function has been demonstrated to increase Glx in the ACC of normal volunteers. The purpose of this study is to determine whether NRX-101, an experimental drug containing a fixed dose combination of D-cycloserine and lurasidone (1) raises Glx by a greater amount than either placebo or lurasidone alone in patients with bipolar depression, and (2) whether that elevation in Glx is correlated with a decrease in depression.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. 18 to 65 years of age, inclusive, at screening.
2. Able to understand and provide written and dated informed consent prior to screening. Deemed likely to comply with study protocol and communicate AEs and other clinically important information, and agree to be hospitalized to complete screening and initiate experimental treatment.
3. Resides in a stable living situation, in the opinion of the investigator
4. Has an identified reliable informant, in the opinion of the investigator
5. Diagnosed with bipolar disorder (BD) according to the criteria defined in the DSM-5. The diagnosis of BD will be made by a psychiatrist and supported by the MINI 7.0.2.
6. Suicidal ideation or behavior as evidenced by an answer of "Yes" to item 2 or item 3 on the C-SSRS.
7. A score of greater than or equal to 20 on the MADRS.
8. In good general health, as ascertained by medical history, physical examination (including measurement of seated vital signs), clinical laboratory evaluations, and electrocardiogram
9. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized [status post hysterectomy, bilateral tubal ligation], or post-menopausal with last menses at least one year prior to screening); or
   2. Childbearing potential, and meets the following criteria:

   i. Using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or sexually abstinent.

   ii. Negative urinary pregnancy test at screening, confirmed by a second negative urinary pregnancy test at randomization prior to receiving study treatment.

   iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and pre-ketamine baseline.
10. Body mass index between 18-35kg/m2.
11. Concurrent psychotherapy will be allowed if the type and frequency of the therapy (e.g., weekly or monthly) has been stable for at least three months prior to screening and is expected to remain stable for the duration of the study.
12. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, or trazodone) will be allowed if the therapy has been stable for at least four weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study. Subjects can also continue treatment with benzodiazepines used for anxiety if therapy has been stable for at least four weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female who is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or before oral dosing of investigational product.
4. Current DSM-5 diagnosis of moderate or severe substance use disorder (except marijuana or tobacco use disorder) within the 12 months prior to screening. Substance abuse cannot be the precipitant of entry to treatment.
5. Subjects with a lifetime history of PCP/ketamine drug use, or failed use of ketamine for depression.
6. History of schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.
7. History of anorexia nervosa, bulimia nervosa, or eating disorder NOS (OSFED) within five years of screening.
8. Has dementia, delirium, amnestic, or any other cognitive disorder.
9. Any major psychiatric disorder, including a personality disorder, which is clinically predominant to BD at screening, or has been the primary focus of treatment predominant to BD at any time within six months prior to screening.
10. Current major psychiatric disorder, diagnosed at screening with the MINI 7.0.2, that is the primary focus of treatment, with BD as the secondary focus of treatment, within the past six months.
11. A clinically significant abnormality on the screening physical examination that might affect safety or study participation, or that might confound interpretation of study results according to the study clinician.
12. Current episode of:

    1. Untreated hypertension, (Stage 1 or greater) as defined by a systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at screening on two of three measurements at least 15 minutes apart. If untreated due to missing medication dose/s this is not exclusionary.
    2. Hypertension, Stage 2, as defined by a systolic blood pressure ≥155 mmHg or diastolic blood pressure ≥99 mmHg within 1.5 hours prior to ketamine infusion on two of three measurements at least 15 minutes apart at the pre-ketamine assessment (on Day 0 at Visit 1).
    3. Recent myocardial infarction (within one year).
    4. Syncopal event within the past year.
    5. Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2.
    6. Angina pectoris.
    7. Heart rate <50 or >105 beats per minute at screening, pre-ketamine infusion (Day 0) or at randomization (Day 1).
    8. QTcF ≥450 msec at screening for men, ≥ 470 msec for women, pre-ketamine infusion (Day 0), or at randomization (Day 1), on two of three measurements at least 15 minutes apart.
13. History of hypertension, or on antihypertensives for the purpose of lowering blood pressure, with either an increase in antihypertensive dose or increase in the number of antihypertensive drugs used to treat hypertension over the last two months.
14. Chronic lung disease, excluding asthma.
15. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the screening clinician, is deemed associated with significant injury to or malfunction of the CNS; or history of significant head trauma within the past two years.
16. Presents with any of the following lab abnormalities:

    a. Subjects with diabetes mellitus fulfilling any of the following criteria: i. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.0 % at screening.

    ii. Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.

    iii. Not under physician care for diabetes mellitus. iv. Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the four weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than eight weeks.

    b. Any other clinically significant abnormal laboratory result (as determined by the investigator and medical monitor) at the time of the screening.
17. Any current or past history of any physical condition which, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation.
18. Subjects on exclusionary concomitant psychotropic medications (see Appendix 1) as defined in the study manual.
19. At randomization, subjects prescribed more than one agent in each category;

    1. Approved antidepressants (e.g., SSRIs, SNRIs, TeCAs, fluoxetine), but not 5-HT-2a antagonists (lurasidone, aripiprazole, olanzapine, quetiapine)
    2. Mood stabilizers (e.g., lithium, carbamazepine, valproic acid)
20. Subjects with exclusionary laboratory values (see Table 2).
21. Known allergies to lurasidone or Latuda, cycloserine or Seromycin, or the excipients mannitol, croscarmellose sodium, magnesium stearate, silicon dioxide, and/or HPMC (hydroxypropylmethylcellulose).
22. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
23. Study site personnel and/or persons employed by NeuroRx, Inc. or Target Health or by the investigator or study site (i.e., permanent, temporary contract worker, or designee responsible for the conduct of the study), or an immediate family member (i.e., spouse or parent, child, or sibling [biological or legally adopted]) of such persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Glx | Immediate
  Mean change in Glx Area Under the Curve (AUC) measured in 15 minute increments over 2 hours at following experimental drug vs. comparator

SECONDARY OUTCOMES:
Depression | 4 weeks
  Depression as measured by score on the Montgomery Asberg Depression Rating Scale (MADRS). The MADRS is a 10 item scale with each item scored from 0 (best) to 6 (worst) for a total possible score of 60.
Suicidal ideation (1) | 4 weeks
  Suicidal ideation as measured on the Columbia Suicidal Severity Rating Scale (C-SSRS) cored from 0 to 5,
Suicidal ideation (2) | 6 hours
  Suicidal ideation as measured by item 10 of the Montgomery Asberg Depression Rating Scale (scored from 0 "best" to 6 "worst")

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T Kantrowicz, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dong Z, Grunebaum MF, Lan MJ, Wagner V, Choo TH, Milak MS, Sobeih T, Mann JJ, Kantrowitz JT. Relationship of Brain Glutamate Response to D-Cycloserine and Lurasidone to Antidepressant Response in Bipolar Depression: A Pilot Study. Front Psychiatry. 2021 Jun 2;12:653026. doi: 10.3389/fpsyt.2021.653026. eCollection 2021. PMID 34149476
- [Result] Milak MS, Rashid R, Dong Z, Kegeles LS, Grunebaum MF, Ogden RT, Lin X, Mulhern ST, Suckow RF, Cooper TB, Keilp JG, Mao X, Shungu DC, Mann JJ. Assessment of Relationship of Ketamine Dose With Magnetic Resonance Spectroscopy of Glx and GABA Responses in Adults With Major Depression: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2013211. doi: 10.1001/jamanetworkopen.2020.13211. PMID 32785636
- See also: FDA Biomarker Letter of Support — https://www.fda.gov/media/112706/download
- See also: Listing of FDA biomarker qualification programs — https://www.fda.gov/drugs/biomarker-qualification-program/letter-support-los-initiative